CLINICAL TRIAL: NCT00527007
Title: Impact of External Cooling in Septic Shock Patients
Brief Title: External Cooling in Septic Shock Patients
Acronym: sepsis-cool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Saliha DJANE, Department of Clinical Research of Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCR06012
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2008-08

CONDITIONS: Septic Shock
Keywords: Vasopressor; Epinephrine; Norepinephrine; Cooling; Fever; ICU
MeSH Terms: conditions — Shock, Septic; Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Other: External cooling
- B (No Intervention)

INTERVENTIONS:
Other: External cooling — External cooling
  Arms: A

SUMMARY:
The rapidity of the resolution of cardiovascular failure has a strong impact on septic shock patients' outcome. The aim of this multicenter randomized controlled trial is to determine whether external cooling might accelerate improvement in cardiovascular function.

DETAILED DESCRIPTION:
Patients suffering from septic shock need fluid resuscitation and vasopressor therapy for restoring cardiovascular function. Corticosteroids and activated protein C have been both proposed for vascular tone improvement. While external cooling is largely used in ICU febrile patients, benefits and risks of fever treatment during sepsis have been rarely studied. Surveys show that external cooling is usual care applied by nurses themselves without medical order.

The control of thermal balance might decrease cardiac output and oxygen consumption, and reduce serum lactate concentration. However some animal studies have suggested that fever might be essential for host defence. This trial compares two strategies of fever management on vasopressor dependence in septic shock patients. In the treatment group, external cooling is applied to normalize the body temperature between 36°5 C and 37°C, while control patients receive any fever treatment. The goal for mean arterial pressure is the same in the two groups and vasopressor withdrawal is determined by similar algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Documented or suspected infection
* Body temperature > 38.3°C
* Persistent hypotension despite fluid resuscitation and need for vasopressor infusion to maintain mean arterial pressure > 65 mmHg.
* Invasive mechanical ventilation
* Intravenous sedation

Exclusion Criteria:

* Temperature > 41°C
* Age < 18 years
* Pregnancy
* Continuous renal replacement therapy
* Paracetamol or NSAI administration within 6 hours before inclusion
* Need for paracetamol and/or NSAI therapy during the study period
* Burns or Lyell syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with a decrease in the dose of vasopressors of 50% 48 hours after enrolment | 48 hours after enrolment

SECONDARY OUTCOMES:
Maximal dose of vasopressors | within 48 hours after enrolment
SOFA score evolution | on Day 3, Day 7, Day 14
Number of vasopressor free days in the ICU | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Frederique SCHORTGEN, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Schortgen F, Charles-Nelson A, Bouadma L, Bizouard G, Brochard L, Katsahian S. Respective impact of lowering body temperature and heart rate on mortality in septic shock: mediation analysis of a randomized trial. Intensive Care Med. 2015 Oct;41(10):1800-8. doi: 10.1007/s00134-015-3987-7. Epub 2015 Jul 23. PMID 26202042